CLINICAL TRIAL: NCT05866588
Title: The Effect Of Nursing Care Based On The Transitional Theory Of Meleis On Primiparous Women's Mothering Role Performance and Parent Self-Efficient
Brief Title: The Effect of Nursing Care on Maternal Role Performance and Parental Self-Efficacy of Primiparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ebru Özcan, lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EOzcan
Record Dates: First submitted 2023-05-01; First posted 2023-05-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Primiparous Women
Keywords: Primiparity; Self Efficacy; Mothers; Parenting
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Experimental Design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participants in the experimental group will receive training and counseling consisting of a total of 8 modules from the 28th week of pregnancy to the fourth month of the postpartum period.
  Interventions: Behavioral: Physical, psychological and spiritual nursing care (Nursing Therapeutics)
- Control group (No Intervention): No educational counseling will be applied to the women in the control group. These participants will receive routine antenatal, natal and postnatal care

INTERVENTIONS:
Behavioral: Physical, psychological and spiritual nursing care (Nursing Therapeutics) — 1. Follow-up: To make a presentation about the physiological and psychological changes during pregnancy. do dream work
  2. Follow-up: Providing education and counseling for childbirth.
  3. Follow-up: Training and role rehearsal on mother-infant interaction, breastfeeding and infant care.
  4. Follow-up: To provide counseling on the issues needed with the approaching of the birth.
  5. Follow-up: Teaching about conscious parenting and mother-infant, father-infant interaction.
  6. Tracking. To provide education, counseling and social support on the other roles of the mother in life such as wife role, working woman role, social role.
  7. Follow-up: To evaluate the transition to motherhood.
  8. Follow-up: To evaluate the outcomes of transition to motherhood and adjustment to motherhood according to expected completion time.
  Arms: experimental group

SUMMARY:
Being a mother is a major and developmental life event involving the transition from an existing and known reality to a new unknown reality, in which the woman gains a new role. In the literature, factors such as age, social support, physical and psychosocial well-being, unrealistic positive or negative expectations, and readiness for the role of mother have been stated that affect maternal identity development, maternal self-efficacy and motherhood role performance. In addition, it has been emphasized that some women are especially at risk in this process. Primiparous (first time giving birth) women are among the groups at risk. Being a first-time mother is an important developmental transition in life, and change is an inevitable element of this process. A prompt and sensitive assessment of my antenatal and postnatal needs and appropriate planning of care are key to effectively supporting women in the transition to motherhood. Therefore, it is thought that individualized nursing care based on Transition theory will be a useful conceptual framework for primary women to realize a healthy transition to motherhood. No research has been found in the literature that evaluates the maternal role performance and parental self-efficacy of primiparous women based on a theory. In this direction, it is thought that this study will shed light on the planning of nursing care to be offered during the transition to motherhood, contribute to the nursing literature, women can make a healthy transition to the role of motherhood, and the risks such as unhealthy transition, role inadequacy, adverse effects on mother and baby health will be minimized. The aim of this study is to determine the Effect of Nursing Care Based on Meleis' Transition Theory on the Maternal Role Performance and Parental Self-Efficacy of Primiparous Women.

DETAILED DESCRIPTION:
Being a mother is a major and developmental life event that includes the transition from an existing and known reality to a new unknown reality, in which the woman gains a new role. Acquiring the role of motherhood; The development of maternal identity is a transformational transition process that includes women's trust in their interactions with their babies, feeling competent as a mother, internalizing the role of motherhood, and integrating the role of motherhood into other existing roles in life. Transition has been defined as moving from one state, condition or place to another. Transitions involve movement from one state of mind to another that develops over time. While individuals, families or societies experience unfamiliar environments and emotions during transitions, they face uncertainty about what they may experience in the post-transition period.

During the transition to motherhood, women may experience unrealistic positive or negative prenatal expectations, disruptions in their daily lives and routines. As a result of these, it will be inevitable that health and well-being will be negatively affected in this process. While especially negative experiences, insufficient social support, unreliable information, negative criticism and attitudes from the environment, stress, anxiety and depression, and generalized care away from individuality negatively affect the development of motherhood identity, readiness for the role of motherhood, having sufficient information, having social support. Factors such as getting professional support, high self-esteem of the mother also affect the development of motherhood identity and motherhood role performance positively. Schumacher and Meleis reported that mothers adapt more to their post-transition roles with a positive transition period and maternal identity acquisition. At the same time, maternal identity development helps the mother to cope with and manage her negative emotions, to feel empowered and free, and positively affects the psychosocial development of women. In the transition to motherhood, the woman's satisfaction from the role of mother and the feeling of self-sufficiency as a mother are the basic components for the acquisition of the motherhood role. Maternal role acquisition has a significant impact on the quality of parenting behavior and the infant's mental development. Motherhood requires women to combine their previous roles with the parenting role after becoming a mother. Being satisfied with the role of motherhood, mother-infant interaction and healthy transition process together with attachment contribute to the acquisition of a flexible and adaptable identity. In other words, maternal role satisfaction has a great role in adapting to the mother's roles in marriage, work, family, spouse's family and social life, as well as motherhood. Studies have shown that being satisfied with the role of mother and an effective mother-infant interaction with the acquisition of motherhood identity positively affect the cognitive and motor development stages of children, their problem-solving skills and psychosocial development. In another study, it was determined that babies who do not communicate effectively with their mothers and cannot bond securely with their mothers experience social isolation during childhood and adolescence. Mercer stated that a woman's self-confidence in the role of mother and feeling competent as a parent are important in reaching the identity of motherhood. In other words, a healthy transition to motherhood is also affected by mothers' beliefs in their competence to be parents. Knowing how to fulfill a role is insufficient for successful role performance. The individual also needs a sense of competence. Parental efficacy has two important components: self-efficacy and satisfaction. Self-efficacy is a cognitive process in which an individual evaluates their ability to cope with or overcome different situations. Parental self-efficacy is defined as "parents' expectations regarding their ability to parent successfully and a parent's sense of being able to positively influence their child's behavior and development". Negative thoughts and concerns in the process of becoming a mother negatively affect women's parental self-efficacy. The higher the perception of self-efficacy, the more likely the woman is to use new skills, especially when a situation becomes difficult.

In the literature, factors such as age, social support, physical and psychosocial well-being, unrealistic positive or negative expectations, and readiness for the role of mother have been stated that affect maternal identity development, maternal self-efficacy and motherhood role performance. In addition, it has been emphasized that some women are especially at risk in this process. Primiparous (first time giving birth) women are among the groups at risk. Being a first-time mother is an important developmental transition in life, and change is an inevitable element of this process. Studies have shown that in the early postpartum period, primiparous women feel more tired, depressed and have more difficulty in assuming the role of motherhood than multiparous women. In addition, primiparous women have lower maternal role satisfaction and self-efficacy perceptions . Low perceived self-efficacy is a risk factor for antenatal depression. It has also been found that primiparous women feel more fear of labor pain and birth complications and have higher levels of anxiety about the negative attitudes of health professionals. Other difficulties faced by primiparous women during the transition to motherhood in studies include routine care of the baby, inadequacy in infant safety and breastfeeding, increased levels of stress, anxiety and depression, and postpartum functional insufficiency. Qualitative studies focusing on the experiences of primiparous people in the transition to motherhood draw attention to the health care providers who do not spare enough time for themselves and answer their questions, and their dissatisfaction with maternity care, information transfer on baby care and self-care, skills training, and the need for more comprehensive guidance and support from health care professionals.

The transition to motherhood is highly subjective and can be experienced very differently from one woman to another. Therefore, every woman has different physiological and psychological care needs during the transition to motherhood. When these care needs are not met, their physiological and psychological health may be adversely affected. Although nurses are at the center of transition processes, they have a very special position to evaluate the physical and psychosocial needs of individuals who are faced with changes and to provide them with holistic and individual care so that they can complete the transition process in a healthy way. In Meleis' Transition Theory; It has been defined which nursing practices nurses can use so that individuals in transition can experience healthy transitions. According to Meleis, by taking the transition theory as a guide, nurses understand the level of awareness of the individual, the responsibilities to be taken, the change to be experienced, the start and expected end time of the transition, the critical turning points, the impact of the change on daily life, the stages the individual goes through and their reactions at different stages of this process. they care for the individual in this direction. Rapid and sensitive assessment of my prenatal and postnatal needs and appropriate planning of care are key to effectively supporting women in transition to motherhood. Therefore, it is thought that individualized nursing care based on Transition theory will be a useful conceptual framework for primary women to realize a healthy transition to motherhood. No research has been found in the literature that evaluates the maternal role performance and parental self-efficacy of primiparous women based on a theory. In this direction, it is thought that this study will shed light on the planning of nursing care to be offered during the transition to motherhood, contribute to the nursing literature, women can make a healthy transition to the role of motherhood, and the risks such as unhealthy transition, role inadequacy, adverse effects on mother and baby health will be minimized.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the research voluntarily.
* To be able to read and write Turkish.
* Not to have a diagnosed psychiatric disease or communication problem.
* Having a mobile phone capable of receiving and playing video messages.
* Being healthy and having a single pregnancy.
* To be between 28-32 weeks of pregnancy.
* Living with a spouse or partner.

Exclusion Criteria:

* Not accepting to participate in the research voluntarily.
* Not being literate in Turkish.
* Having a diagnosed psychiatric illness or communication problem.
* Lack of mobile phone capable of receiving and playing video messages.
* Having a high-risk or multiple pregnancy.
* Being under 28 weeks or over 32 weeks pregnant.
* Not living with a spouse or partner.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
The Scale of Being the Structure of a New Baby | It is applied to both groups on the 7th postpartum day.
  With the Maternity Role Performance, women's evaluation of their motherhood experiences, their satisfaction with the motherhood role and their perception of life changes will be evaluated.
  The measurement is made to reveal the qualitative aspects of the mother related to being the mother of a new baby. The score distribution of the scale is between 17-153. It has 2 sub-dimensions. Each sub-dimension is evaluated within itself.
The Scale of Being the Structure of a New Baby | It is applied to both groups on the 1th month.
  With the Maternity Role Performance, women's evaluation of their motherhood experiences, their satisfaction with the motherhood role and their perception of life changes will be evaluated.
  The measurement is made to reveal the qualitative aspects of the mother related to being the mother of a new baby. The score distribution of the scale is between 17-153. It has 2 sub-dimensions. Each sub-dimension is evaluated within itself.
The Scale of Being the Structure of a New Baby | It is applied to both groups on the 4th month.
  With the Maternity Role Performance, women's evaluation of their motherhood experiences, their satisfaction with the motherhood role and their perception of life changes will be evaluated.
  The measurement is made to reveal the qualitative aspects of the mother related to being the mother of a new baby. The score distribution of the scale is between 17-153. It has 2 sub-dimensions. Each sub-dimension is evaluated within itself.
Parental Self-Efficacy Scale | It is applied to both groups on the 4th month.
  With Parental Self-Efficacy, it will be evaluated whether women feel competent in the role of mother.
  It was developed to determine the personal judgments of new parents with their first and only 3-6 month old babies regarding their competencies in the parent role. There are sub-dimensions of Meeting Needs, Parental Competence, Relief of Discomfort, Coping with Illness and Social Interaction. As the score obtained from the scale increases, self-efficacy increases.

SECONDARY OUTCOMES:
Edinburgh Postpartum Depression Scale | Measurements are made at 28 weeks of gestation for both groups.
  The scale can be used to determine the risk of depression. The scale consists of 10 items in total. The total score is calculated by assigning a value between 0 and 3 for each item. The cut-off score of the scale for screening was calculated as 12.
Edinburgh Postpartum Depression Scale | Measurements are made at 38 weeks of gestation for both groups.
  The scale can be used to determine the risk of depression. The scale consists of 10 items in total. The total score is calculated by assigning a value between 0 and 3 for each item. The cut-off score of the scale for screening was calculated as 12.
Edinburgh Postpartum Depression Scale | Measurements are made at 7th postpartum day for both groups.
  The scale can be used to determine the risk of depression. The scale consists of 10 items in total. The total score is calculated by assigning a value between 0 and 3 for each item. The cut-off score of the scale for screening was calculated as 12.
Edinburgh Postpartum Depression Scale | Measurements are made at 1th postpartum month for both groups.
  The scale can be used to determine the risk of depression. The scale consists of 10 items in total. The total score is calculated by assigning a value between 0 and 3 for each item. The cut-off score of the scale for screening was calculated as 12.
Edinburgh Postpartum Depression Scale | Measurements are made at 4th postpartum month for both groups.
  The scale can be used to determine the risk of depression. The scale consists of 10 items in total. The total score is calculated by assigning a value between 0 and 3 for each item. The cut-off score of the scale for screening was calculated as 12.
Prenatal Maternity Expectations Scale | For each group, measurements are made at the 28th gestational week of pregnancy.
  It measures prenatal maternal expectations. A total score ranging from 34 to 170 is also obtained from the scale. Accordingly, a high score from the scale represents an unrealistic positive expectation, a low score represents an unrealistic negative expectation, while a moderate score represents a realistic expectation.
Prenatal Maternity Expectations Scale | For each group, measurements are made at the 36th gestational week of pregnancy.
  It measures prenatal maternal expectations. A total score ranging from 34 to 170 is also obtained from the scale. Accordingly, a high score from the scale represents an unrealistic positive expectation, a low score represents an unrealistic negative expectation, while a moderate score represents a realistic expectation.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru ÖZCAN, Study Director — Ondokuz Mayıs University
Locations (1):
- Kastamonu Provincial Health Directorate, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of the research will be shared with third parties with the research report when the research is concluded and published. If the editor wishes to see the raw data during publication, it will be forwarded to him.
Supporting Information: CSR
Time Frame: Data available after research is published
Access Criteria: The research can be accessed according to the journal in which it was published.

REFERENCES:
- [Result] Mercer RT. Becoming a mother versus maternal role attainment. J Nurs Scholarsh. 2004;36(3):226-32. doi: 10.1111/j.1547-5069.2004.04042.x. PMID 15495491
- [Result] Mercer RT, Walker LO. A review of nursing interventions to foster becoming a mother. J Obstet Gynecol Neonatal Nurs. 2006 Sep-Oct;35(5):568-82. doi: 10.1111/j.1552-6909.2006.00080.x. PMID 16958712
- [Result] Schumacher KL, Meleis AI. Transitions: a central concept in nursing. Image J Nurs Sch. 1994 Summer;26(2):119-27. doi: 10.1111/j.1547-5069.1994.tb00929.x. PMID 8063317
- [Result] SmithBattle L, Freed P. Teen Mothers' Mental Health. MCN Am J Matern Child Nurs. 2016 Jan-Feb;41(1):31-6; quiz E3-4. doi: 10.1097/NMC.0000000000000198. PMID 26474475
- [Result] Barimani M, Vikstrom A, Rosander M, Forslund Frykedal K, Berlin A. Facilitating and inhibiting factors in transition to parenthood - ways in which health professionals can support parents. Scand J Caring Sci. 2017 Sep;31(3):537-546. doi: 10.1111/scs.12367. Epub 2017 Jan 31. PMID 28144992
- [Result] Bassi M, Delle Fave A, Cetin I, Melchiorri E, Pozzo M, Vescovelli F, Ruini C. Psychological well-being and depression from pregnancy to postpartum among primiparous and multiparous women. J Reprod Infant Psychol. 2017 Apr;35(2):183-195. doi: 10.1080/02646838.2017.1290222. Epub 2017 Feb 19. PMID 29517362
- [Result] Tsai SS, Wang HH. Role changes in primiparous women during 'doing the month' period. Midwifery. 2019 Jul;74:6-13. doi: 10.1016/j.midw.2019.03.007. Epub 2019 Mar 18. PMID 30908975
- [Derived] Ozcan E, Temiz S. The impact of nursing care based on transition theory on maternal role performance and parental self-efficacy in primiparous women: a randomized controlled study. BMC Nurs. 2025 Apr 5;24(1):377. doi: 10.1186/s12912-025-03054-4. PMID 40188345